CLINICAL TRIAL: NCT03875040
Title: Is There a Relationship Between Kinesiophobia and Physical Activity Level in Patients With Knee Osteoarthritis?
Brief Title: Knee Osteoarthritis, Kinesiophobia and Physical Activity
Status: Completed | Type: Observational
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dr. Melek Aykut Selçuk, Principal investigator, Aksaray University Training and Research Hospital
Other Study IDs: 2018/67
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Fear of Pain; Knee Osteoarthritis; Physical Activity
Keywords: kinesiophobia; osteoarthritis; fear of movement; tampa; physical inactivity
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity; Kinesiophobia; Osteoarthritis; Sedentary Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: kinesiophobia — patients who have a high-level or low-level kinesiophobia have been evaluated.

SUMMARY:
Although the importance of regular physical activity in patients with knee osteoarthritis is known, and fear of movement is considered as one of the causes of physical inactivity and is widely researched in terms of its role in the pathogenesis of pain, there remains to be limited number of studies on kinesiophobia in these patients. In this study, we aimed to evaluate the levels of kinesiophobia and physical activity in patients with knee osteoarthritis and to investigate whether they were associated with demographic characteristics, body mass index, pain intensity, depression, disability, radiological grade, and quality of life.

DETAILED DESCRIPTION:
A total of 96 female and male patients aged 50 to 75 years with knee osteoarthritis (OA) and knee pain lasting for more than three months (knee pain intensity over 20 mm on Visual Analog Scale-VAS) were included in the study. The severity of pain at night, pain at rest and activity-related pain was evaluated by Visual Analog Scale (VAS), kinesiophobia by Tampa Scale of Kinesiophobia (TSK) and Brief Fear of Movement Scale (BFOM), depression by the Beck Depression Inventory (BDI), disability by the Western Ontario and McMaster Universities Arthritis Index (WOMAC), physical activity level by the International Physical Activity Questionnaire (IPAQ) short form and quality of life by the Short Form 12 Health Survey Questionnaire (SF-12). Age, gender, marital status, educational status, additional disease, drug history, and sociodemographic data such as BMI were obtained from the patients and recorded in the evaluation form.

ELIGIBILITY:
Inclusion Criteria:

knee osteoarthritis aged 50 to 75 years knee pain lasting for than three months knee pain intensity over 20 mm on Visual Analog Scale-VAS

Exclusion Criteria:

knee operation, Malignant diseases Systemic infectious diseases inflammatory diseases Fibromyalgia syndrome physical therapy and/or a knee injection within the last three months antidepressants, pregabalin or duloxetine usage

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients presenting to Aksaray Training and Research Hospital Physical Medicine and Rehabilitation Outpatient Clinic between April 2018 and October 2018, who volunteered to participate in the study and fulfilled the inclusion criteria, completed the questionnaire forms.
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
Tampa Scale of Kinesiophobia | 4-8 minutes
  Based on a four-point Likert type, this scale contains 17 items that evaluate fear and anxiety related to physical activity. A total score of greater than 37 is accepted as statistically significant and interpreted as a high level of kinesiophobia. Minimal and maximal scores could be between 17-68 points. Higher scores indicate higher levels of kinesiophobia.
International Physical Activity Questionnaire Short Form | 5-10 minutes
  This questionnaire consists of seven items that measure the duration of the participants' physical activity, walking and sitting within the last seven days in the metabolic equivalent (MET)-min/week unit. 3 or more days of vigorous activity of at least 20 minutes per day or 5 or more days of moderate-intensity activity and/or walking of at least 30 minutes per day or 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 600 MET-minutes/week are proposed to be moderate level. Vigorous-intensity activity on at least 3 days and accumulating at least 1500 MET-minutes/week or 7 or more days of any combination of walking, moderate- or vigorous-intensity activities accumulating at least 3000 MET-minutes/week are proposed to be high level.Some activity is reported but not enough to meet categories of moderate or high levels, it is proposed to be low level.
Beck Depression Inventory | 10 minutes
  This is a 21-item questionnaire that investigates the characteristic attitudes and symptoms of depression. A score of 10 or higher indicates depression. Minimal and maximal scores can be 0-63 points. Higher scores indicate higher levels of depression.
Visual Analog Scale for the Evaluation of Pain | 0.5 minutes
  For this evaluation, the patient is asked to mark his/her severity of pain on a horizontal 10-cm line with number 0 on one end representing "no pain" and number 10 on the other end indicating "very severe pain". Higher scores indicate higher levels of pain intensity.
Short Form-12 Health Survey Questionnaire | 5 minutes
  A scale used to evaluate the quality of life, consisting of 12 items inquiring general health, physical condition, physical limitations, mental status, social status, pain, energy and mental limitation over a total score of 100 points. SF-12 is an abbreviated version of SF-36 and has been proven to be reliable and valid. In this study, we evaluated the patients' total, physical and mental SF-12 scores
Western Ontario and McMaster Universities Arthritis Index | 10 minutes
  A 24-item measure that was developed to evaluate pain, joint stiffness and physical functions in individuals with knee and hip OA. A higher score indicates a higher level of pain, stiffness and functional limitation. In our study, we used the WOMAC total score.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Aykut Selçuk, Principal Investigator — Ankara Akyurt Public Hospital
Locations (1):
- Aksaray Training and Research Hospital, Aksaray, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunn AH, Schwartz TA, Arbeeva LS, Callahan LF, Golightly Y, Goode A, Hill CH, Huffman K, Iversen MD, Pathak A, Taylor SS, Allen KD. Fear of Movement and Associated Factors Among Adults With Symptomatic Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2017 Dec;69(12):1826-1833. doi: 10.1002/acr.23226. Epub 2017 Nov 6. PMID 28371481
- [Background] Shelby RA, Somers TJ, Keefe FJ, DeVellis BM, Patterson C, Renner JB, Jordan JM. Brief Fear of Movement Scale for osteoarthritis. Arthritis Care Res (Hoboken). 2012 Jun;64(6):862-71. doi: 10.1002/acr.21626. Epub 2012 Jan 30. PMID 22290689

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT03875040/Prot_SAP_000.pdf